CLINICAL TRIAL: NCT05419102
Title: Retrospective Study of Implants With Peri-implantitis Surgically Treated Using Enamel Matrix Derivative (EMD)
Status: Completed | Type: Observational
Sponsor: North Dallas Dental Health (Other)
Responsible Party: Principal Investigator, Thomas G Wilson, Jr. DDS, Private Practitioner, North Dallas Dental Health
Other Study IDs: EMD Implant 1
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Determination of Beneficial Effect of Using Enamel Matrix Derivative During Implant Treatment
Keywords: dental implant; peri-implantitis; enamel matrix derivative
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: peri-implantitis surgery with enamel matrix derivative — surgical procedures around dental implants with peri-implantits to remove infectious material and apply enamel matrix derivative to the implant.

SUMMARY:
The existing records of a private practice limited to the practice of periodontology were reviewed to locate patients who had been diagnosed with peri-implantitis (failing dental implant) and had been surgically treated utilizing enamel matrix derivative (Commercially available FDA product Emdogain sold by Straumann USA). Various clinical factors were gathered from the existing records. Some of the factors recorded were: retention of the implant, presence of bleeding, presence of further damage, and presence of inflammation. All patients had signed an informed consent for treatment and the anonymous use of their data for research purposes. All HIPA requirements were followed.

DETAILED DESCRIPTION:
See brief summary.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients of record who presented with existing peri-implantitis that was clinically deemed treatable (the implant was not considered hopeless.)

Exclusion Criteria:

* none except for routine medical contraindications for periodontal surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine adult patients in a private periodontal practice.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
retention of the implant | 0.71 to 6.4 years
  Determine if the implant was still present at the time of reevaluation

SECONDARY OUTCOMES:
record the clinical condition of the implant at the time of reevaluation | 0.71 to 6.4 years
  Multiple standard measurements of the clinical condition of the implant were recorded at the time of reevaluation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Wilson, Principal Investigator
Locations (1):
- North Dallas Dental Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No